CLINICAL TRIAL: NCT04562480
Title: A Phase II Study of Hypofractionated Pre-Operative Radiation Therapy for Localized, Resectable Soft Tissue Sarcoma of the Extremity and Superficial Trunk
Brief Title: Radiation Therapy Before Surgery for Localized, Resectable Soft Tissue Sarcoma of the Extremity and Superficial Trunk
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MC1973; NCI-2020-06811 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); MC1973 (Other: Mayo Clinic in Rochester); 19-011871 (Other: Mayo Clinic Institutional Review Board)
Record Dates: First submitted 2020-09-18; First posted 2020-09-24 (Actual); Results first posted 2026-01-16 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2026-01

CONDITIONS: Resectable Soft Tissue Sarcoma; Stage I Soft Tissue Sarcoma of the Trunk and Extremities AJCC v8; Stage IA Soft Tissue Sarcoma of the Trunk and Extremities AJCC v8; Stage IB Soft Tissue Sarcoma of the Trunk and Extremities AJCC v8; Stage II Soft Tissue Sarcoma of the Trunk and Extremities AJCC v8
MeSH Terms: interventions — Radiation Dose Hypofractionation; Radiation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Treatment (hypofractionated radiation therapy, resection) (Experimental): Patients undergo hypofractionated radiation therapy QD (except weekends and holidays) over 3 weeks for a total of 15 fractions. Within 3-6 weeks after completion of radiation therapy, patients undergo surgical resection.
  Interventions: Radiation: Hypofractionated Radiation Therapy; Other: Quality-of-Life Assessment; Other: Questionnaire Administration; Procedure: Resection

INTERVENTIONS:
Radiation: Hypofractionated Radiation Therapy — Undergo hypofractionated radiation therapy
  Other Names: Hypofractionated; Hypofractionated Radiotherapy; hypofractionation; Radiation, Hypofractionated
Other: Quality-of-Life Assessment — Ancillary studies
  Other Names: Quality of Life Assessment
Other: Questionnaire Administration — Ancillary studies
Procedure: Resection — Undergo surgical resection
  Other Names: Surgical Resection

SUMMARY:
This phase II trial investigates the effects of hypofractionated radiation therapy before surgery on wound complications associated with surgery in treating patients with soft tissue sarcoma of the extremity (arms, hands, legs or feet) and superficial trunk that has not spread to other parts of the body (localized) and can be removed by surgery (resectable). Hypofractionated is a shorter radiation therapy treatment length (fewer radiation treatment days) and administers the total radiation dose as larger daily doses, compared to conventionally fractionated therapy.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To report the major acute wound complication rate associated with hypofractionated preoperative radiation therapy, 42.75 Gy in 15 fractions.

SECONDARY OBJECTIVES:

I. To report the 5-year local failure rate associated with hypofractionated preoperative radiation therapy, 42.75 Gy in 15 fractions.

II. To report the 5-year disease-free survival rate associated with hypofractionated preoperative radiation therapy, 42.75 Gy in 15 fractions.

III. To report the 5-year overall survival rate associated with hypofractionated preoperative radiation therapy, 42.75 Gy in 15 fractions.

IV. To report long-term toxicity rates associated with hypofractionated preoperative radiation therapy, 42.75 Gy in 15 fractions.

V. To describe patterns of relapse associated with hypofractionated preoperative radiation therapy, 42.75 Gy in 15 fractions.

VI. To describe patient reported outcomes/quality-of-life outcomes with hypofractionated preoperative radiation therapy, 42.75 Gy in 15 fractions.

OUTLINE:

Patients undergo hypofractionated radiation therapy once daily (QD) (except weekends and holidays) over 3 weeks for a total of 15 fractions. Within 3-6 weeks after completion of radiation therapy, patients undergo surgical resection.

After completion of study treatment, patients are followed up at 4-8 weeks, every 3-4 months for years 1-2, and every 6 months for years 3-5.

ELIGIBILITY:
Inclusion Criteria:

* Newly diagnosed, histological confirmation of soft tissue sarcoma of the extremities (including limb girdle) or superficial trunk that present as either -

  * Deemed a candidate for complete macroscopic resection of the primary sarcoma OR
  * Having had non-oncologic excisional procedure with positive or uncertain resection margins and still be eligible if the evaluating sarcoma surgeon recommends oncologic re-resection of the surgical bed to obtain negative margins after a course of preoperative radiation therapy
* No evidence of nodal or distant metastases as determined by clinical examination on any form of imaging
* Eastern Cooperative Oncology Group (ECOG) performance status (PS) =< 3
* Life expectancy greater than 6 months
* Patients capable of childbearing must use adequate contraception
* Ability to complete questionnaire(s) by themselves or with assistance
* Ability to provide written informed consent
* Willing to return to enrolling institution for follow-up (during the Active Monitoring Phase of the study)

Exclusion Criteria:

* Previous radiation therapy to the site of the sarcoma or area surrounding it such that it would be encompassed by the radiation field needed to treat the current sarcoma. In other words, treatment on this trial would require re-irradiation of tissues
* Patients with nodal or distant metastases
* Rhabdomyosarcoma, soft tissue osteosarcoma, soft tissue Ewing sarcoma, and benign histologies
* Any of the following:

  * Pregnant women
  * Nursing women
  * Men or women of childbearing potential who are unwilling to employ adequate contraception

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2020-11-30 (Actual); Primary Completion 2024-10-31 (Actual); Study Completion 2029-10-31 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Safia K. Ahmed, M.D., Principal Investigator — Mayo Clinic
Locations (3):
- United States (3):
  - Mayo Clinic in Arizona, Scottsdale, Arizona
  - Mayo Clinic in Florida, Jacksonville, Florida
  - Mayo Clinic in Rochester, Rochester, Minnesota

REFERENCES:
- [Result] Ahmed SK, Xu-Welliver M, Dorr M, Steinert KO, Houdek MT, Rose PS, Karim SM, Ashman JB, Goulding KA, Siontis BL, Haddock MG, Petersen IA. Hypofractionated Preoperative Radiation Therapy for Extremity and Superficial Trunk Soft Tissue Sarcomas: Results of a Prospective, Phase 2 Trial. Int J Radiat Oncol Biol Phys. 2025 Nov 15;123(4):980-989. doi: 10.1016/j.ijrobp.2025.05.006. Epub 2025 May 17. PMID 40389098
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Treatment (Hypofractionated Radiation Therapy, Resection)
Started | 120
Completed | 119
Not Completed | 1
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Arm/Group | Treatment (Hypofractionated Radiation Therapy, Resection)
Number analyzed (Participants) | 119
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 63.8 [48.0 to 71.8]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 63
  Male | 56
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 6
  Not Hispanic or Latino | 108
  Unknown or Not Reported | 5
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1
  Asian | 4
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 106
  More than one race | 0
  Unknown or Not Reported | 7
Region of Enrollment [Number; unit: participants]
  United States | 119

OUTCOME MEASURES:

1. Primary Outcome: Major Wound Complications
Description: Will be assessed by the number of patients who experience major wound complications within 120 days following surgery. Major wound complication is defined as secondary unplanned operation under general or regional anesthesia for wound repair (e.g., debridement, operative drainage, or secondary wound closure including rotationplasty, free flaps or skin grafts); or wound management without secondary operation including invasive procedures (e.g., aspiration of seroma or readmission for wound care such as intravenous antibiotics or persistent deep packing for 120 days or longer).
Time Frame: Within 120 days of surgical resection of soft tissue sarcoma following preoperative radiation therapy
Population: Two patients treated with radiation therapy came off study before surgery because of death.
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (Hypofractionated Radiation Therapy, Resection)
Number analyzed (Participants) | 117
Participants
  No | 90
  Yes | 27

2. Secondary Outcome: Local Failure Rate
Description: Defined as any radiographic or pathologic evidence of recurrent disease inside the clinical target volume (CTV) and/ or to within 3 cm from the edge of the CTV. Local failure rate at 5 years (LFR5) will be evaluated by the number of patients free of local failure/recurrence at 5 years.
Time Frame: Up to 1 year
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (Hypofractionated Radiation Therapy, Resection)
Number analyzed (Participants) | 119
Participants | 2

3. Secondary Outcome: Percent Probability of Disease-free Survival at 1 Year
Description: Defined as the time from registration to the earliest date of documentation of local recurrence, regional recurrence, distant recurrence, or death due to any cause
Time Frame: up to 1 year
Measure: Number (95% Confidence Interval); unit: Percent Probability
Groups:
- Treatment (Hypofractionated Radiation Therapy, Resection): Patients undergo hypofractionated radiation therapy QD (except weekends and holidays) over 3 weeks for a total of 15 fractions. Within 3-6 weeks after completion of radiation therapy, patients undergo surgical resection.
  >
  > Hypofractionated Radiation Therapy: Undergo hypofractionated radiation therapy
  >
  > Quality-of-Life Assessment: Ancillary studies
  >
  > Questionnaire Administration: Ancillary studies
  >
  > Resection: Undergo surgical resection
Arm/Group | Treatment (Hypofractionated Radiation Therapy, Resection)
Number analyzed (Participants) | 117
Percent Probability | 86 [79.7 to 92.9]

4. Secondary Outcome: Percent Probability of Overall Survival at 1 Year
Description: Defined as the time from registration date to death due to any cause
Time Frame: Up to 1 year
Measure: Number (95% Confidence Interval); unit: Percent Probability
Arm/Group | Treatment (Hypofractionated Radiation Therapy, Resection)
Number analyzed (Participants) | 117
Percent Probability | 97.0 [93.7 to 100]

5. Secondary Outcome: Incidence of Late Adverse Events
Description: The descriptions and grading scales found in the revised National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) version 5.0 will be utilized for adverse event reporting. The rate of >= grade 2 late adverse events will be estimated by the number of patients with a >= grade 2 late adverse events.
Time Frame: Between 3 months and 24 months after completion of hypofractionated preoperative radiation therapy
Reporting Status: Not Posted

6. Secondary Outcome: Pattern of Relapse
Description: Pattern of relapse will be evaluated by number of patients with patterns of tumor recurrence such as local recurrence, marginal recurrence, regional recurrence, distant metastasis, and second primary tumor.
Time Frame: Up to 1 years
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (Hypofractionated Radiation Therapy, Resection)
Number analyzed (Participants) | 119
Participants | 2

7. Secondary Outcome: Incidence of Adverse Events
Description: The descriptions and grading scales found in the revised NCI CTCAE version 5.0 will be utilized for adverse event reporting. The maximum grade for each type of adverse event will be recorded for each patient, and frequency tables will be reviewed to determine patterns.
Time Frame: Up to 1 year
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (Hypofractionated Radiation Therapy, Resection)
Number analyzed (Participants) | 117
Participants
  Grade 3 | 16
  Grade 4 | 0
  Grade 5 | 1

8. Secondary Outcome: Change in Quality of Life - PROMIS-10
Description: Results from the ten-item Patient Reported Outcomes Measurement Information System (PROMIS-10) questionnaire will be used to evaluate physical and mental health separately. The PROMIS-10 consists of ten items that measure physical health, physical functioning, general mental health, emotional distress, satisfaction with social activities and relationships, ability to carry out usual social activities and roles, pain, fatigue and overall quality of life.
Time Frame: Baseline up to 24 months post-surgery
Reporting Status: Not Posted

9. Secondary Outcome: Change in Quality of Life - TESS
Description: Results from the Toronto Extremity Salvage Score (TESS) questionnaire will be used to evaluate functional outcomes. The TESS was designed as a measure of the difficulty patients have performing routine daily activities. It consists of 31 items with responses from 1 (impossible to do) to 5 (not at all difficult).
Time Frame: Baseline up to 24 months post-surgery
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Up to 1 year
Arm/Group | Treatment (Hypofractionated Radiation Therapy, Resection)
All-Cause Mortality (participants affected / at risk) | 2/117
Serious Adverse Events (participants affected / at risk) | 49/117
Other Adverse Events (participants affected / at risk) | 117/117
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Hypofractionated Radiation Therapy, Resection) (N=117)
Anemia (Blood and lymphatic system disorders) | 1 (2)
Nausea (Gastrointestinal disorders) | 2 (2)
Death NOS (General disorders) | 1 (1)
Fatigue (General disorders) | 11 (12)
Localized edema (General disorders) | 1 (1)
Lung infection (Infections and infestations) | 1 (1)
Skin infection (Infections and infestations) | 1 (1)
Joint range of motion decreased (Musculoskeletal and connective tissue disorders) | 21 (36)
Tumor pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 15 (18)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 1 (1)
Lymphedema (Vascular disorders) | 7 (12)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Hypofractionated Radiation Therapy, Resection) (N=117)
Anal stenosis (Gastrointestinal disorders) | 2 (2)
Anal ulcer (Gastrointestinal disorders) | 2 (2)
Colonic perforation (Gastrointestinal disorders) | 2 (2)
Colonic stenosis (Gastrointestinal disorders) | 2 (2)
Colonic ulcer (Gastrointestinal disorders) | 2 (2)
Diarrhea (Gastrointestinal disorders) | 1 (1)
Duodenal perforation (Gastrointestinal disorders) | 2 (2)
Duodenal stenosis (Gastrointestinal disorders) | 2 (2)
Duodenal ulcer (Gastrointestinal disorders) | 2 (2)
Enterovesical fistula (Gastrointestinal disorders) | 2 (2)
Gastric perforation (Gastrointestinal disorders) | 2 (2)
Gastric stenosis (Gastrointestinal disorders) | 2 (2)
Gastric ulcer (Gastrointestinal disorders) | 2 (2)
Ileal fistula (Gastrointestinal disorders) | 2 (2)
Ileal perforation (Gastrointestinal disorders) | 2 (2)
Ileal stenosis (Gastrointestinal disorders) | 2 (2)
Ileal ulcer (Gastrointestinal disorders) | 2 (2)
Jejunal fistula (Gastrointestinal disorders) | 2 (2)
Jejunal perforation (Gastrointestinal disorders) | 2 (2)
Jejunal stenosis (Gastrointestinal disorders) | 2 (2)
Jejunal ulcer (Gastrointestinal disorders) | 2 (2)
Nausea (Gastrointestinal disorders) | 3 (4)
Rectal fistula (Gastrointestinal disorders) | 2 (2)
Rectal perforation (Gastrointestinal disorders) | 2 (2)
Rectal stenosis (Gastrointestinal disorders) | 2 (2)
Rectal ulcer (Gastrointestinal disorders) | 2 (2)
Small intestinal perforation (Gastrointestinal disorders) | 2 (2)
Small intestinal stenosis (Gastrointestinal disorders) | 2 (2)
Small intestine ulcer (Gastrointestinal disorders) | 2 (2)
Vomiting (Gastrointestinal disorders) | 1 (1)
Edema limbs (General disorders) | 1 (1)
Fatigue (General disorders) | 86 (142)
Localized edema (General disorders) | 53 (129)
Pain (General disorders) | 1 (1)
Sepsis (Infections and infestations) | 1 (1)
Wound infection (Infections and infestations) | 2 (2)
Dermatitis radiation (Injury, poisoning and procedural complications) | 83 (122)
Fracture (Injury, poisoning and procedural complications) | 5 (7)
Fibrosis deep connective tissue (Musculoskeletal and connective tissue disorders) | 50 (137)
Joint range of motion decreased (Musculoskeletal and connective tissue disorders) | 65 (162)
Tumor pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 58 (90)
Bladder perforation (Renal and urinary disorders) | 2 (2)
Urinary fistula (Renal and urinary disorders) | 2 (2)
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 81 (205)
Telangiectasia (Skin and subcutaneous tissue disorders) | 1 (1)
Lymphedema (Vascular disorders) | 29 (74)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2024-04-17): https://cdn.clinicaltrials.gov/large-docs/80/NCT04562480/Prot_SAP_000.pdf
  • Informed Consent Form (2024-06-07): https://cdn.clinicaltrials.gov/large-docs/80/NCT04562480/ICF_001.pdf